CLINICAL TRIAL: NCT03774719
Title: Hand-carried Ultrasound for Ruling Out Hydronephrosis in Acute Kidney Injury and Acute Kidney Disease
Brief Title: Hand-carried Ultrasound to Assess Hydronephrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in staffing, COVID, New US curriculum being developed
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201903192-1985080800
Record Dates: First submitted 2018-12-07; First posted 2018-12-13 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Hydronephrosis; Ultrasound; Acute Kidney Injury
MeSH Terms: conditions — Hydronephrosis; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hand-carried ultrasound arm (Experimental): This is the only arm of the study. It will be comprised of 154 inpatients who had a renal ultrasound ordered or performed within the past 4 hours. The intervention will be performing hand-carried ultrasound to evaluate for presence and degree of hydronephrosis.
  Interventions: Device: Hand-carried ultrasound

INTERVENTIONS:
Device: Hand-carried ultrasound — Hand-carried ultrasound of both kidneys to detect the presence or absence of hydronephrosis. Device used will be the lumify portable ultrasound equipped with the C5-2 curved array transducer (Philips, USA).
  Other Names: Point of care ultrasound; POCUS

SUMMARY:
This study evaluates if trainees can accurately rule out dilation of the renal collecting system on ultrasound (hydronephrosis) using hand-carried ultrasound (HCU). Trainees will undergo a short ultrasound training program. Patients will be adults that are hospitalized and have acute or subacute kidney dysfunction. The investigators will assess sensitivity, specificity, positive and negative predictive value of HCU compared to radiology performed ultrasound, and calculate potential cost savings to the patient and to the healthcare system.

DETAILED DESCRIPTION:
Hand-carried ultrasound is an increasingly popular imaging modality and is widely used by emergency physicians, intensivists, trauma doctors and cardiologists. Renal ultrasonography is commonly ordered for patients with acute kidney injury, with a main focus on identifying obstruction of the collecting system, a rare but potentially reversible cause of acute kidney injury.

This study's aim is to evaluate if nephrology and internal medicine trainees can accurately rule out dilation of the renal collecting system on ultrasound (hydronephrosis) using hand-carried ultrasound (HCU). Trainees will undergo a short, uniform and well described ultrasound training program. Patients will be adults that are hospitalized and have acute or subacute kidney dysfunction. The investigators will assess sensitivity, specificity, positive and negative predictive value of HCU compared to radiology performed ultrasound, and calculate potential cost savings to the patient and to the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* Inpatient admission to Barnes Jewish Hospital (BJH)
* Patient has a diagnosis of Acute kidney injury (AKI) or Acute kidney Disease (AKD)
* Renal ultrasound ordered or performed within the past 4 hours

Exclusion Criteria:

* End-stage renal disease
* History of kidney transplant
* Stable chronic kidney disease
* Current diagnosis of renal cell carcinoma
* Pregnant women
* Morbid obesity (BMI >40)
* Rash or active skin lesions overlying the scanning area (left or right flank)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited after presenting to the hospital between May 2019 and April 2023. First participant was enrolled May 6, 2019 and last participant enrolled May 24, 2019.
Pre-assignment Details: 18 patients were screened, 6 met inclusion criteria, agreed to participate and were enrolled in the study.
Groups:
- Hand-carried Ultrasound Arm: This is the only arm of the study. It will include inpatients who had a renal ultrasound ordered or performed within the past 4 hours. The intervention will be performing hand-carried ultrasound to evaluate for presence and degree of hydronephrosis.
  Hand-carried ultrasound: Hand-carried ultrasound of both kidneys to detect the presence or absence of hydronephrosis. Device used will be the lumify portable ultrasound equipped with the C5-2 curved array transducer (Philips, USA).
Period: Overall Study
Arm/Group | Hand-carried Ultrasound Arm
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hand-carried Ultrasound Arm
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 65.5 [60 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Absence of Hydronephrosis
Description: The number of participants for whom none of the kidneys imaged with hand-carried ultrasound have hydronephrosis (dilation of the collecting system) is reported
Time Frame: Through study completion, up to an average of 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Hand-carried Ultrasound Arm
Number analyzed (Participants) | 6
Participants | 4

2. Secondary Outcome: Direct Costs of Hand-carried Ultrasound
Description: Direct costs in $ of hand-carried ultrasound will be calculated and compared to the costs of radiology performed ultrasound. For hand-carried ultrasound, this will include costs of purchasing the device, training costs, yearly depreciation of the hand-carried ultrasound device. For radiology performed ultrasound, this will include the sonographer's fee, radiologist fee for interpretation of the result, transportation fee by hospital transport and depreciation of the ultrasound machine.
Time Frame: Through study completion, up to an average of 1 day
Population: Data regarding costs were not collected by research team at the time of the study.
Arm/Group | Hand-carried Ultrasound Arm
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Ultrasound Image Quality
Description: Ultrasound image quality assessed by a blinded independent radiologist. The quality will be deemed either excellent, good, fair or poor by the radiologist.
Time Frame: Through study completion, up to an average of 1 day
Population: Data regarding image quality was not collected by research team at the time of the study.
Arm/Group | Hand-carried Ultrasound Arm
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Technical Difficulty of the Ultrasound Study
Description: How technically difficult was it for the trainees to obtain the images (patient intubated, obesity etc.) as graded by the trainees who performed the ultrasound scans themselves. Trainees will grade difficulty using the following measurement scale (1) Technically easy: trainee able to get clear images of both kidneys within a timeframe of 10 minutes (2) Technically challenging: Trainee able to get clear images of kidneys but requiring more than 10 minutes of scanning time (3) Technically difficult: trainee unable to get clear images of both kidneys independent of time spent scanning.
Time Frame: Through study completion, up to an average of 1 day
Population: Data regarding technical difficulty of the study was not collected by the research team.
Arm/Group | Hand-carried Ultrasound Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Time from start of ultrasound evaluation to end of ultrasound evaluation, up to 2 hours
Arm/Group | Hand-carried Ultrasound Arm
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Single center, study terminated did not reach enrollment target due to change in PI and COVID pandemic. No statistical analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT03774719/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT03774719/ICF_002.pdf